CLINICAL TRIAL: NCT06849440
Title: The Effect of Childbirth Preparation Education on Perceived Stress and Traumatic Birth Perception in Pregnant Women
Brief Title: Effectiveness of Childbirth Preparation Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Antalya Bilim University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-101
Record Dates: First submitted 2025-01-14; First posted 2025-02-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-02

CONDITIONS: Perception of Traumatic Birth; Perceived Stress
Keywords: childbirth; childbirth preparation; percieved stress; perception of traumatic birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Training group (Experimental): The sociodemographic data collection form and the perceived stress and traumatic birth perception scales as pre-tests will be applied to the pregnant women who accept the study before the childbirth training. After the pre-test, the pregnant women will be given face-to-face childbirth preparation training in a classroom environment during four sessions. When the participants complete the training sessions, the scales will be applied as a post-test. The data collection process will be completed after the application of the scales.
  Interventions: Behavioral: Training

INTERVENTIONS:
Behavioral: Training — Participants will be divided into groups of ten and the training is planned in 4 sessions. Session contents are prepared as sharing general information on preparation for birth, explanation of frequently applied interventions in labor, explanation of non-drug pain relieving methods, teaching and practicing active birth positions that help the labor progress. The duration of the sessions is planned as 2 hours on average.

SUMMARY:
The act of birth, which is considered a natural event, is an act that the mother will remember with positive experiences in her life if it progresses normally. However, sometimes birth can be perceived as stressful and traumatic for women. Stress during pregnancy is a problem that should be emphasized and managed due to its negative effects on the health of the mother and the baby. As the pregnancy progresses, the levels of stress hormones may increase. In addition, the thought of spontaneous birth exposes women to physical discomfort, stress and uncertainty during pregnancy. The perception of traumatic birth is an important concept that emerges as a result of the woman's mental birth scenario, the information she has acquired about birth, and every situation she experiences during the birth, and also affects the postpartum period. In studies conducted in Turkey using the Traumatic Birth Perception Scale, it was determined that 23.6% and 26.9% of women experienced a high level of traumatic birth perception. Nulliparity, negative feelings about birth, inadequate antenatal care, inadequate psychosocial support, risky pregnancies, and lack of information about birth are among the factors that may cause traumatic birth perception. Physical and mental preparation for birth and information about pain management are considered to be the basic elements of prenatal education classes. There are study results indicating that birth preparation classes benefit women in many aspects such as self-sufficiency, reduced fear of birth, and positive pregnancy experience. No study results have been found in the literature examining the effect of birth preparation education on the perception of traumatic birth during pregnancy. Based on this, this study was needed to examine the effect of pregnant women's participation in childbirth preparation training on their perceived stress level and perception of traumatic birth.

ELIGIBILITY:
28-34th weeks of pregnancy Agree to participate in the study Be literate Be able to speak and understand Turkish

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-05-09 (Actual); Study Completion 2025-05-09 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale (PSS) | Pre-test and immediately post-test
  It was developed by Cohen et al. (1983). The scale was adapted to Turkish by Eskin et al. (2013). The PSS, which consists of 14 items in total, was designed to measure the degree to which a number of situations in a person's life are perceived as stressful. Participants evaluate each item on a 5-point Likert-type scale ranging from "Never (0)" to "Very often (4)". 7 of the items containing positive expressions are scored reversely. Scores vary between 0 and 56. A high score indicates a high perception of stress. In the study by Eskin et al., the Cronbach's alpha value of the scale was found to be 0.84.

SECONDARY OUTCOMES:
Traumatic Birth Perception Scale (TBPS) | Pre-test and immediately post-test
  The Traumatic Birth Perception Scale (TBPS) was developed by Yalnız et al. (2016) to determine the perception of traumatic birth, and its validity and reliability studies were conducted. The original study was conducted on women aged 18-40. The final version of the scale consists of 13 items. Each item is in the form of an ordinal scale and is scored between 1 (lowest score) and 10 (highest score). The scores obtained from each item are added together. As the score obtained from the scale increases, it shows that the level of perception of birth as traumatic increases. The score obtained from the scale varies between 0 and 130. According to the total score of the scale; 0-26 points indicate "very low", 27-52 points indicate "low", 53-78 points indicate "medium", 79-104 points indicate "high", and 105-130 points indicate "very high" level of perception of traumatic birth. The Cronbach alpha value was found to be 0.89 in the original study of the scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Antalya Bilim University, Antalya, Turkey (Türkiye)